CLINICAL TRIAL: NCT00104156
Title: Qigong Therapy for Osteoarthritis at Knees
Brief Title: Qigong Therapy for Individuals With Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT001352-01A2 (NIH)
Record Dates: First submitted 2005-02-23; First posted 2005-02-24 (Estimated); Last update posted 2008-01-25 (Estimated); Status verified 2008-01

CONDITIONS: Osteoarthritis
Keywords: Knee pain; Arthritis; Qigong; Qi; Meditation; Breathing Exercises
MeSH Terms: conditions — Osteoarthritis; Arthritis

INTERVENTIONS:
Procedure: External Qigong therapy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Qigong therapy, an ancient Chinese practice, for pain relief and symptom improvement in people with knee osteoarthritis (OA).

Study hypotheses: 1) Qigong therapy will result in greater reduction of pain and greater symptom improvement than sham treatment. 2) Individuals with a history of complementary and alternative medicine (CAM) use will be more likely to experience benefits of Qigong therapy than those without such experience.

DETAILED DESCRIPTION:
OA is the leading cause of disability in the United States. Standard treatment for OA is drug therapy; however, cost, side effects, and varying levels of effectiveness warrant the need for development of new treatments. Qigong therapy, which involves deep meditation, breathing exercises, and the harnessing of energy, may be an effective treatment for OA.

According to traditional Chinese medicine, Qi (Chi) is the "life force" that flows through the body and keeps people healthy and vital. In the practice of traditional Chinese medicine, arthritis is thought to be due to a blockage of the flow of Qi or a buildup of abnormal or damaging Qi. It is believed that releasing this buildup or breaking the blockage of Qi through Qigong therapy may relieve OA symptoms.

Participants will be randomly assigned to receive five sessions of either Qigong therapy or sham treatment over a period of 2 weeks. During Qigong therapy, a therapist will send his or her Qi to the arthritic knees through touch and meditation. Similar body work will be performed during the sham treatment, but no Qi will be harnessed. Self-report scales that measure pain, stiffness, anxiety, daily drug use, CAM use, and overall functioning will be used to assess participants. The assessments will occur at study start and at a 3-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteoarthritis at least 6 months prior to study entry
* Able to understand English

Exclusion Criteria:

* Inflammatory joint disease affecting leg movement
* Knee replacement surgery on the OA knee
* Depo-corticosteroid knee injections within 3 months prior to study entry
* Pain in hips or lower back affecting leg movement
* New arthritis drugs or other painkillers within 2 weeks prior to study entry
* Investigational drugs within 30 days prior to study entry
* Asthma requiring oral corticosteroids within 4 weeks prior to study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Pain, stiffness, and physical function scale results

SECONDARY OUTCOMES:
McGill Pain Questionnaire (MPQ-SF) results
Spielberger State-Trait Anxiety Scale (STAI) results
Daily dosage of drugs for pain relief
Range of motion for knees
Time to walk 50 feet

CONTACTS AND LOCATIONS:
Overall Officials: Kevin W. Chen, PhD MPH, Principal Investigator — Division of Addiction Psychiatry, University of Medicine and Dentistry, New Jersey-Robert Wood Johnson Medical School; Leonard Sigal, MD, Principal Investigator — Rheumatology Department - Biomedical Sciences Program, University of Medicine and Dentistry, New Jersey-Robert Wood Johnson Medical School
Locations (2):
- United States (2):
  - University of Medicine and Dentistry, New Jersey-Robert Wood Johnson Medical School, Newark, New Jersey
  - University of Medicine and Dentistry, New Jersey-Robert Wood Johnson Medical School, Piscataway, New Jersey